CLINICAL TRIAL: NCT00290030
Title: A Double-Blind Randomized Parallel Group Study of Alfuzosin 10mg OD Versus Placebo in the Management of Acute Urinary Retention in Patients With a First Episode Due to Benign Prostatic Hyperplasia (BPH)
Brief Title: ALFAURUS : A DB Randomized Parallel Group Study of Alfuzosin 10mg OD vs Placebo in the Management of AUR in Patients With a 1st Episode Due to BPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4428; SL 770499-10
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Prostatic Hyperplasia; Acute Urinary Retention
Keywords: acute urinary retention; International Prostate Symptom Score (IPSS)
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
To assess the efficacy of alfuzosin 10mg OD in the management of acute urinary retention associated with BPH.

To assess the safety of alfuzosin in this population and health care consumption.

DETAILED DESCRIPTION:
Double-blind, placebo controlled, randomized Multicenter, Phase III study comparing 2 parallel groups (alfuzosin 10mg OD or placebo) in patients with a first episode of acute urinary retention related to BPH.The acute episode is managed with catheterization and with study drug treatment for 2 to 3 days, followed by an active voiding trial to assess the patients' ability to void after catheter removal.

Those patients who successfully void will continue their randomized treatment for a total treatment duration of 6 months. For all patients who are prematurely withdrawn during the study, a post-study (clinic or phone) visit will be performed for collection of health care consumption data.

ELIGIBILITY:
Inclusion Criteria:

* Male aged over 50 years
* Having given his written consent
* Presenting with a first episode of painful acute urinary retention related to BPH
* With a catheterized urine volume between mL and mL at the time of retention

Exclusion Criteria:

* Associated urological diseases / troubles (e.g. infection or surgery of prostate, urinary retention f neurogenic origin
* Iatrogenic causes of urinary retention

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2001-05; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Successful voiding in initial period (using an active voiding trial)
No relapse during the 6 month treatment period
No need / indication for surgery during the initial or 6 month treatment periods

SECONDARY OUTCOMES:
To assess the safety of alfuzosin in this population, and health care consumption

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi

REFERENCES:
- See also: Related Info — http://www.sanofi-aventis.com